CLINICAL TRIAL: NCT04318951
Title: Impact of Intensive Social Interaction on Post-Stroke Depression in Individuals With Aphasia
Acronym: CONNECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BB 033/17
Record Dates: First submitted 2020-03-17; First posted 2020-03-24 (Actual); Results first posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Post-stroke Depression; Post-stroke Aphasia
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive communicative-pragmatic social interaction. (Experimental): Intensive Language-Action Therapy (ILAT).
  Interventions: Behavioral: Intensive communicative-pragmatic social interaction.; Behavioral: Standard care.
- Standard care. (Other): All participants will receive standard care.
  Interventions: Behavioral: Standard care.

INTERVENTIONS:
Behavioral: Intensive communicative-pragmatic social interaction. — ILAT requires individuals with aphasia to engage in social interaction. Groups of three patients and a therapist are seated around a table and provided with picture cards showing different objects (e.g., bottle). Each card has a duplicate that is owned by one of the other players. The goal is to obtain this duplicate from a fellow player by requesting the depicted object (e.g., "Give me the […]"). If the duplicate is available, the addressee hands over the corresponding card to the person who initiated the request sequence. If the duplicate is not available, the addressee rejects the request. In the event of misunderstandings, the players ask clarifying questions. Throughout the training, participants use formulaic expressions to indicate whether a request is accepted ("Here you are," "Thank you," "You're welcome"), rejected ("I'm sorry," "No problem," "Too bad") or unclear ("Pardon me?"). Treatment duration will be four weeks.
  Arms: Intensive communicative-pragmatic social interaction.
Behavioral: Standard care. — Depending on the participants' diagnoses and needs, standard care will include: occupational therapy (2-3 hours of weekly practice), physiotherapy (3 hours of weekly practice), and speech-language therapy (2-3 hours of weekly practice with non-communicative, impairment-specific exercises). Standard care will be delivered in accordance with state-of-the-art procedures in rehabilitation centers certified in Germany. Treatment duration will be four weeks.

SUMMARY:
The present parallel-group, single-center, blinded-assessment controlled trial seeks to explore the feasibility - in terms of high completion rates - and potential efficacy of intensive communicative-pragmatic social interaction for treatment of post stroke depression in subacute aphasia. Apart from evidence of treatment feasibility, the primary hypothesis predicts significantly greater progress on self-report and clinician-rated measures of depression severity after (i) intensive communicative-pragmatic social interaction combined with standard care, compared to (ii) standard care alone.

DETAILED DESCRIPTION:
Background. Individuals with post-stroke aphasia often experience a profound loss of abilities to engage in social interaction, one major reason for increased risk of depression after a cerebrovascular accident. Impaired communication skills in aphasia can prevent classical forms of psychotherapy, thus emphasizing the need for new rehabilitation strategies alongside antidepressant medication.

Aims. The present parallel-group, single-center, blinded-assessment controlled trial seeks to explore the feasibility - in terms of high completion rates (primary outcome) - and potential efficacy (co-primary and secondary outcomes, as defined below) of intensive communicative-pragmatic social interaction for treatment of post-stroke depression in subacute aphasia. In this early time window after a cerebrovascular accident, prevalence of post-stroke depression is generally high.

Methods. Treatment is based on a linguistically validated protocol that encourages individuals with aphasia to use neural resources of verbal communication embedded in intensive social interaction. In a routine-healthcare outpatient setting, 60 individuals with post-stroke depression and subacute aphasia will be assigned to one of two groups in a pseudorandomized fashion: (i) intensive communicative-pragmatic social interaction combined with standard care, or (ii) standard care alone.

Endpoints and Outcomes. Apart from evidence of treatment feasibility, endpoint will be change on self-report and clinician-rated measures of depression severity (co-primary outcomes: Beck's Depression Inventory, BDI; and Hamilton Rating Scale for Depression, HAM-D) after a 1-month treatment period (5 hours of weekly training). Secondary outcomes include measures evaluating self-efficacy, quality of life, and language performance (secondary outcomes: Self-Efficacy Questionnaire; and Aachen Aphasia Test, AAT).

Hypotheses. Aside from evidence of treatment feasibility, the primary hypothesis predicts significant between-group differences on BDI and HAM-D scores, indicating greater reduction in depression severity with intensive communicative-pragmatic social interaction over and above standard care alone. Secondary analyses will focus on the Self-Efficacy Questionnaire as an external criterion to explore the psychometric adequacy of the self-report co-primary outcome, the BDI, and consider progress in language performance from onset to end of treatment on the AAT to account for the potential relationship between change in cognitive-affective distress and verbal expression skills.

Clinical Relevance. The current proof-of-concept trial will investigate the feasibility and potential efficacy of intensive communicative-pragmatic social interaction as a means to promote recovery from post-stroke depression in subacute aphasia. The results obtained will determine the design of a subsequent phase-III randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Left-hemisphere cortical or subcortical stroke;
* Native speaker of German;
* Right-handedness according to the Edinburgh Handedness Inventory (Oldfield, 1971);
* Diagnosis of post-stroke depression, as defined in the International Statistical Classification of Diseases and Related Health Problems (ICD-11);
* Diagnosis of aphasia, as confirmed by standardized tests (e.g., Huber et al., 1984); and
* Late subacute or consolidation phase (i.e., 0.5-6 months following stroke) where risk of post-stroke depression is particularly high (Shi et al., 2014).

Exclusion Criteria:

* Other neurological conditions;
* Pre-morbid history of depression;
* Other psychopathological conditions;
* Severely impaired vision or hearing that may prevent participants from engaging in intensive communicative-pragmatic social interaction during therapy or testing, thus adopting routine-healthcare standards from a large-scale phase-III randomized controlled trial (Breitenstein et al., 2017);
* Serious non-verbal cognitive deficits; and
* No informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Stahl, PhD, Principal Investigator — University Medicine of Greifswald & Medical School Berlin; Agnes Flöel, MD, Principal Investigator — University Medicine of Greifswald
Locations (1):
- MEDIAN-Klinik Berlin-Kladow, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stahl B, Van Lancker Sidtis D. Tapping into neural resources of communication: formulaic language in aphasia therapy. Front Psychol. 2015 Oct 20;6:1526. doi: 10.3389/fpsyg.2015.01526. eCollection 2015. No abstract available. PMID 26539131
- [Background] Stahl B, Mohr B, Dreyer FR, Lucchese G, Pulvermuller F. Using language for social interaction: Communication mechanisms promote recovery from chronic non-fluent aphasia. Cortex. 2016 Dec;85:90-99. doi: 10.1016/j.cortex.2016.09.021. Epub 2016 Oct 15. PMID 27842269
- [Background] Stahl B, Mohr B, Buscher V, Dreyer FR, Lucchese G, Pulvermuller F. Efficacy of intensive aphasia therapy in patients with chronic stroke: a randomised controlled trial. J Neurol Neurosurg Psychiatry. 2018 Jun;89(6):586-592. doi: 10.1136/jnnp-2017-315962. Epub 2017 Dec 22. PMID 29273692
- [Background] Breitenstein C, Grewe T, Floel A, Ziegler W, Springer L, Martus P, Huber W, Willmes K, Ringelstein EB, Haeusler KG, Abel S, Glindemann R, Domahs F, Regenbrecht F, Schlenck KJ, Thomas M, Obrig H, de Langen E, Rocker R, Wigbers F, Ruhmkorf C, Hempen I, List J, Baumgaertner A; FCET2EC study group. Intensive speech and language therapy in patients with chronic aphasia after stroke: a randomised, open-label, blinded-endpoint, controlled trial in a health-care setting. Lancet. 2017 Apr 15;389(10078):1528-1538. doi: 10.1016/S0140-6736(17)30067-3. Epub 2017 Mar 1. PMID 28256356
- [Background] Huber W, Poeck K, Willmes K. The Aachen Aphasia Test. Adv Neurol. 1984;42:291-303. No abstract available. PMID 6209953
- [Background] Oldfield RC. The assessment and analysis of handedness: the Edinburgh inventory. Neuropsychologia. 1971 Mar;9(1):97-113. doi: 10.1016/0028-3932(71)90067-4. No abstract available. PMID 5146491
- [Background] Shi YZ, Xiang YT, Wu SL, Zhang N, Zhou J, Bai Y, Wang S, Wang YL, Zhao XQ, Ungvari GS, Chiu HF, Wang YJ, Wang CX. The relationship between frontal lobe lesions, course of post-stroke depression, and 1-year prognosis in patients with first-ever ischemic stroke. PLoS One. 2014 Jul 8;9(7):e100456. doi: 10.1371/journal.pone.0100456. eCollection 2014. PMID 25003990
- [Result] Stahl B, Millrose S, Denzler P, Lucchese G, Jacobi F, Floel A. Intensive Social Interaction for Treatment of Poststroke Depression in Subacute Aphasia: The CONNECT Trial. Stroke. 2022 Dec;53(12):3530-3537. doi: 10.1161/STROKEAHA.122.039995. Epub 2022 Sep 20. PMID 36124755
- See also: Documentary feature on the present clinical trial. — http://www.cbs.mpg.de/podcast/leben-nach-schlaganfall.mp3

RESULTS

PARTICIPANT FLOW:
Groups:
- Intensive Communicative-pragmatic Social Interaction.: Intensive Language-Action Therapy (ILAT).
  Intensive communicative-pragmatic social interaction: ILAT requires individuals with aphasia to engage in social interaction.
Period: Overall Study
Arm/Group | Intensive Communicative-pragmatic Social Interaction. | Standard Care.
Started | 30 (1 March 2020) | 30 (1 March 2020)
Completed | 30 (15 January 2022) | 30 (15 January 2022)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: BDI and HAM-D.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive Communicative-pragmatic Social Interaction. | Standard Care. | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (11.8) | 74.7 (10.9) | 72.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 38
  Male | 13 | 9 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 30 | 30 | 60
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 30 | 30 | 60
BDI. [Mean (Standard Deviation); unit: units on a scale] — Beck's Depression Inventory. Scale range: 0-120. Higher values represent higher degree of depression.
  units on a scale | 28.2 (6.2) | 24.0 (3.4) | 26.1 (14.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Beck's Depression Inventory, BDI.
Description: This self-report measure of depression severity is derived from a standardized questionnaire known for its good psychometric properties, including construct validity and test-retest reliability, in individuals without aphasia. Scale range: 0-120. Higher values represent higher degree of depression.
Time Frame: Change from 1 day before start of treatment until immediately after 4 weeks of treatment.
Population: Post-Stroke Depression and Subacute Aphasia
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intensive Communicative-pragmatic Social Interaction. | Standard Care.
Number analyzed (Participants) | 30 | 30
score on a scale | -12.6 [-17.5 to -7.7] | -5.8 [-11.7 to -2.6]

2. Primary Outcome: Change in Hamilton Rating Scale for Depression, HAM-D. Higher Values Represent Higher Degree of Depression.
Description: This clinician-rated measure of depression severity is known for its good psychometric properties, including construct validity and test-retest reliability, in individuals without aphasia. Scale range: 0-35.
Time Frame: Change from 1 day before start of treatment until immediately after 4 weeks of treatment.
Population: Post-Stroke Depression and Subacute Aphasia
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intensive Communicative-pragmatic Social Interaction. | Standard Care.
Number analyzed (Participants) | 30 | 30
score on a scale | -5.0 [-6.4 to -3.6] | -3.3 [-4.5 to -2.1]

3. Secondary Outcome: Self-Efficacy Questionnaire.
Description: This self-report questionnaire was conceived to quantify a person's confidence to overcome obstacles encountered when completing a difficult task. Results are expressed on a Likert scale ranging from 0 (very low self-efficacy) to 3 (very high self-efficacy). Results are expressed as sum scores ranging from 0 (very low self-efficacy) to 30 (very high self-efficacy). Reduced self-efficacy is discussed as one risk factor for depression. This instrument was used only for cross-sectional assessment, not for longitudinal assessment, to serve as an external criterion to explore the psychometric adequacy of the self-report co-primary outcome, the BDI.
Time Frame: Immediately after 4 weeks of treatment (used only as an external criterion to explore the psychometric adequacy of the self-report co-primary outcome, the BDI)
Population: Post-Stroke Depression and Subacute Aphasia
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intensive Communicative-pragmatic Social Interaction. | Standard Care.
Number analyzed (Participants) | 30 | 30
score on a scale | 20.1 (7.1) | 18.3 (7.8)

4. Other Pre Specified Outcome: Change in Aachen Aphasia Test, AAT.
Description: This standardized aphasia test battery was found to be sensitive to treatment-induced short-term progress in language performance. To address the potential relationship between changes in cognitive-affective distress and verbal expression skills, we will use the combined AAT subscales "Repetition" and "Naming" as a covariate in exploratory evaluations. The AAT subscales "Repetition" and "Naming" as well as the resulting combined average score are based on a T-score distribution (M = 50; SD = 10). Higher T-scores represent better verbal expression skills. The results below indicate change over time.
Time Frame: Change from 1 day before start of treatment until immediately after 4 weeks of treatment.
Population: Post-Stroke Depression and Subacute Aphasia
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Intensive Communicative-pragmatic Social Interaction. | Standard Care.
Number analyzed (Participants) | 30 | 30
T-score | 3.5 [2.0 to 5.0] | 2.9 [1.0 to 4.8]

ADVERSE EVENTS:
Time Frame: 3 weeks
Description: Behavioral intervention; no risk expected.
Arm/Group | Intensive Communicative-pragmatic Social Interaction. | Standard Care.
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT04318951/Prot_SAP_000.pdf